CLINICAL TRIAL: NCT05593367
Title: Effects of Vitamin D on Gut Microbiota, Intestinal Barrier in Patients With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: Effects of Vitamin D on Gut Microbiota, Intestinal Barrier in IBS-D Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022014
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: IBS-D; Vitamin D; Gut microbiota; Intestinal barrier;

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal Specimen, Serum Specimen；Intestinal Mucosa Specimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VD-， VD deficiency group: The IBS-D patients whose serum 25(OH)D level was<20ng/ml
- VD+， VD normal group: The IBS-D patients whose serum 25(OH)D level was ≥20ng/ml

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disease. Evidence suggests that the concentration of serum VD is decreased in IBS patients, particularly in IBS-D. After giving a supplementation of VD, some symptoms of these patients were relieved to a certain degree. However, the specific mechanism still remains unclear.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disease, which is due to the gut microbiota disturbances, intestinal mucosal barrier dysfunction, and brain-gut axis dysfunction. Vitamin D (VD), a fat-soluble vitamin, has been found to be associated with gut microbiota, intestinal mucosal barrier and NLRP3 in inflammatory bowel disease, nonalcoholic fatty liver disease and other diseases. The concentration of serum VD is decreased in IBS patients, particularly in IBS-D. And the symptoms of IBS patients seems to be connected with the level of serum VD. After giving a supplementation of VD, some symptoms of these patients were relieved to a certain degree. However, the specific mechanism still remains unclear.We designed a study to figure out the effects of serum VD on gut microbiota, intestinal mucosal barrier and in patients with IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* ①IBS-D patients meeting the Roman IV diagnostic criteria: recurrent abdominal pain, averaging at least 1 day per week in the last 3 months, with 2 or more of the following: associated with defecation, accompanied by changes in defecation frequency, accompanied by changes in fecal properties or appearance. (Symptoms have been present for at least 6 months before diagnosis, and meet the above diagnostic criteria in the last 3 months; >1/4 (25%) stools were Bristol Stool Scale type 6 or 7, and <1/4 (25%) stools were Bristol Stool Scale type 1 or 2); ② The age ranged from 18 to 65.

Exclusion Criteria:

* ① History of other gastrointestinal diseases, such as inflammatory bowel disease, infection, cancer, abdominal radiation or surgery, hepatobiliary and pancreatic diseases; ② Taking vitamin D drugs, calcium, contraceptives, glucocorticoids, probiotics, antibiotics, antidepressants, etc.; ③ Pregnancy and lactation; ④ Diabetes mellitus, thyroid disease, osteoporosis, etc.; ⑤ Complicated with serious heart, liver, lung, kidney, blood, serious mental diseases and other systemic diseases; (6) Boston Intestinal Preparation Scale score <6; The cecum was not detected by endoscopy. ⑦ Unwilling to participate or unable to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBS-D Patients who meet the above criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | 1 week before colonoscopy
  Detect the fecal microbiome by 16S rRNA gene sequencing.
intestinal barrier | During the colonoscopy
  Detect the expressions of Z0-1, occludin in intestinal mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Fei Dai, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided